CLINICAL TRIAL: NCT03293641
Title: The Effects of Zinc Supplementation in Children With Sickle Cell Disease in Western Kenya: a Pilot Study
Brief Title: Zinc Supplementation in Children With Sickle Cell Disease in Western Kenya
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lucas Otieno Tina, MD MSc (Other)
Collaborators: GlaxoSmithKline (Industry); Strathmore University (Other)
Responsible Party: Sponsor-Investigator, Lucas Otieno Tina, MD MSc, Principal Investigator, Kenya Medical Research Institute
Organization: Kenya Medical Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KEMRI SSC 2925
Record Dates: First submitted 2017-04-14; First posted 2017-09-26 (Actual); Last update posted 2017-09-26 (Actual); Status verified 2017-09

CONDITIONS: Sickle Cell Disease; Zinc Deficiency; Infection
Keywords: Children, Sickle Cell Disease, Zinc
MeSH Terms: conditions — Anemia, Sickle Cell; Infections | interventions — Zinc Sulfate; Standard of Care; Folic Acid; Proguanil; Penicillin V; Hydroxyurea

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Pilot Trial in which children aged 6 months to less than 13 years were randomized on a ration of 1:1 to receive the Zinc plus Standard of Care versus Standard of Care Management for Sickle Cell Disease
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zinc Sulfate Tablet (Experimental): Zinc Sulfate Tablet 10 mg, 3 times a week plus Standard of Care for 6 months
  Interventions: Dietary Supplement: Zinc Sulfate Tablets; Drug: Standard of Care
- Control Arm (Placebo Comparator): Standard of Care for 6 months
  Interventions: Drug: Standard of Care

INTERVENTIONS:
Dietary Supplement: Zinc Sulfate Tablets — Zinc Sulfate Tablets 3 times every 7 days for 6 months.
  Other Names: Zincos
  Arms: Zinc Sulfate Tablet
Drug: Standard of Care — Folic Acid, Proguanil, Penicillin V, Hydroxyurea over 6 months
  Other Names: Folic Acid, Proguanil, Penicillin V, Hydroxyurea

SUMMARY:
Zinc is a nutritionally essential trace element found in previous studies to reduce growth retardation and improve immune function, which may also result in decreased incidence of infectious diseases including malaria, pneumonia and diarrhea. Sickle Cell Disease (SCD) patients are known to be susceptible to zinc deficiency and appear to benefit from zinc supplementation. The proposed pilot research project aims to investigate the influence of zinc supplementation on incidence of malaria infections, incidence of bacterial infections and investigate the influence of zinc supplementation on morbidity in children with SCD in western Kenya. The differences in incidence of morbidity and other secondary endpoints will be compared between the zinc group and the control group.

DETAILED DESCRIPTION:
Zinc is a nutritionally essential trace element found in previous studies to reduce growth retardation and improve immune function, which may also result in decreased incidence of infectious diseases including malaria, pneumonia and diarrhea. SCD patients are known to be susceptible to zinc deficiency and appear to benefit from zinc supplementation. Despite these findings, SCD patients in Kenya have not benefited from zinc supplementation programs due to a lack of research and findings to inform policy in the East African-setting. The proposed pilot research project aims to investigate the influence of zinc supplementation on incidence of malaria infections in children with SCD; investigate the influence of zinc supplementation on incidence of bacterial infections (e.g. S pneumoniae, H influenzae and non-typhi Salmonella species) in children with SCD and investigate the influence of zinc supplementation on morbidity in children with SCD in western Kenya. A 6 month randomized controlled pilot trial involving children with SCD aged 6 months to less than 13 years, being treated and followed up routinely at the KEMRI-site and other selected health facilities in Western Kenya for SCD will be enrolled. The children will be randomized into two arms, with the Intervention Group receiving the recommended Ministry of Health (MoH)/World Health Organization (WHO) standard care in addition to three times weekly zinc supplementation (10 mg) and the Control Group receiving standard MoH care alone over a six month period. At baseline, at 3 months and at 6 months, clinical and laboratory evaluations, including serum zinc levels, malaria blood slides, anthropometric measurements and other indicated laboratory tests will be conducted.The differences in incidence of morbidity and other secondary endpoints will be compared between the zinc group and the control group. The results are expected to determine the scientific basis for a larger clinical trial to determine the need for the addition of zinc supplement to the management of sickle cell disease.

ELIGIBILITY:
Inclusion Criteria:

* Male or female infants and children ≥ 6 months and < 13 years of age with confirmed SCD.
* Written informed consent obtained from the participant's parent/Legally Acceptable Representative (LAR).
* Available to participate for the study duration (approximately six months)

Exclusion Criteria:

* Written informed consent NOT obtained from the participant's parent/Legally Acceptable Representative (LAR).
* Profound clinical evidence of current immunosuppression or evidence of active AIDS defining illness i.e. WHO HIV clinical stage III/IV
* History of allergic reactions to zinc or any other ingredients in the supplement
* History of any neurologic disorders or seizures
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic, renal functional abnormality, as determined by physical examination or laboratory screening tests
* Hemoglobin ≤7.0 g/dL in children aged 6 months to ≤ 2 years.
* Hemoglobin ≤ 6 g/dL in children aged >2yrs to <13 years.
* Total White Cell Count below normal range <4.5 x 103/uL
* Use of any investigational or non-registered drugs or vaccines or planned use
* Simultaneous participation in any other clinical trial
* Any other findings that the investigator feels would increase the risk of having an adverse outcome from participation in the trial.

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2016-05-20 (Actual); Primary Completion 2017-01-19 (Actual); Study Completion 2017-01-19 (Actual)

PRIMARY OUTCOMES:
Measurement of change in zinc levels from baseline at study conclusion. | 6 months
  Zinc Levels in Plasma

SECONDARY OUTCOMES:
Number of malaria episodes among recipients of zinc versus controls diagnosed by RDT or Microscopy. | 6 months
  Malaria Incidence
Number of episodes of bacterial infections among recipients of zinc versus controls diagnosed by culture. | 6 months
  Bacterial Infection Incidence
Incidence of malnutrition among recipients of zinc versus controls diagnosed based on anthropometric measurements. | 6 months
  Anthropometric Measurements i.e. Weight, Height and Mid Upper Arm Circumference
Occurrences of Adverse Events (AEs) during the 6 month follow-up period among recipients of zinc versus controls. | 6 months
  Adverse Events including Serious Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Lucas O Tina, MD MSc, Principal Investigator — KEMRI/CREATES, Strathmore University

IPD SHARING:
Plan to Share IPD: No